CLINICAL TRIAL: NCT03276091
Title: Evaluation of a Motivational Phone Call Strategy to Improve Colonoscopy Participation, for Patients With a Positive Immunochemical Fecal Test : Colofit + Study
Brief Title: Colonoscopy Motivation for Patients With Positive Immunochemical Fecal Test
Acronym: Colofit+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Soler-Michel (Other)
Responsible Party: Sponsor-Investigator, Patricia Soler-Michel, ADEMAS69, Association pour le Dépistage Organisé des Cancers dans le Rhône
Organization: Association pour le Dépistage Organisé des Cancers dans le Rhône (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDRCB 2017-A00635-48
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Colon Cancer
Keywords: colonoscopy; immunochemical fecal test; screening
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COLOFIT+ Study (Experimental): Personnalized motivational phone call, done by a medical physician
  Interventions: Behavioral: Colofit+ intervention

INTERVENTIONS:
Behavioral: Colofit+ intervention — Personnalized phone call, done by the medical student in the name of Adémas-69, organized cancers screening in the Rhône area association. This is a motivational call to encourage patients with an immunochemical fecal test positive, to realized their colonoscopy.

SUMMARY:
Patients with an immunochemical fecal test positive, have to undergo a colonoscopy. Around 10% doesn't realize the colonoscopy. This study evaluate the impact of a motivational phone call (given by a doctor) to improve colonoscopy participation. And try to understand why this patients don't want to make this examination.

ELIGIBILITY:
Inclusion Criteria:

* immunochemical fecal test positive but no colonoscopy performed despite a full sequence of reminder (3 letters)

Exclusion Criteria:

* colonoscopy done

Ages: 51 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Participation to the colonoscopy | From date of phone call until the date of first documented colonoscopy assessed up to 6 months
  Colonoscopy done six months after our phone call

SECONDARY OUTCOMES:
reasons for rejecting colonoscopy | Reasons for rejecting colonoscopy will be assessed during the phone call only, and assessed until the end of this phone call
  we will ask to patients why they don't realized their colonoscopy
cancer and adenoma detected | From date of phone call until the date of first documented colonoscopy result assessed up to 6 months after phone call
  number of cancer and adenoma detected during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Ponchon, PHD, Study Director — Hopital Edouard Herriot
Locations (1):
- Ademas-69, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gandilhon C, Soler-Michel P, Vecchiato L, Chaunier C, Fay I, Walter T, Rivory J, Saurin JC, Ponchon T, Pioche M. A motivational phone call improves participation to screening colonoscopy for those with a positive FIT in a national screening programme (NCT 03276091). Dig Liver Dis. 2018 Dec;50(12):1309-1314. doi: 10.1016/j.dld.2018.08.007. Epub 2018 Aug 17. PMID 30197186